CLINICAL TRIAL: NCT06315699
Title: Randomized, Double-blind, Controlled Study of Clomastine Fumarate in the Treatment of Williams Syndrome
Brief Title: Clemastine Fumarate in the Treatment of Neurodevelopmental Delays in Williams Syndrome
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: QL000001; MR-37-24-002019 (Registry Identifier: Chinese Clinical Trial Registry)
Record Dates: First submitted 2024-03-04; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Williams Syndrome; Child; Neurodevelopmental Delay
Keywords: clemastine fumarate; Williams syndrome; MRI
MeSH Terms: conditions — Williams Syndrome | interventions — Clemastine; Fructose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clemastine (Experimental): Clemastine，tablet，0.15mg/kg/d，two months
  Interventions: Drug: Clemastine Fumarate Tablets
- fructose (Placebo Comparator)
  Interventions: Dietary Supplement: fructose

INTERVENTIONS:
Drug: Clemastine Fumarate Tablets — The dose was administered 2mg once daily in a double-blind random crossover method
  Arms: Clemastine
Dietary Supplement: fructose — The dose was administered 2mg once daily in a double-blind random crossover method
  Arms: fructose

SUMMARY:
This study focuses on therapeutic targets for cognitive, motor, and social impairments in Williams syndrome by reversing brain myelin defects caused by GTF2I. The primary objective of the study was to test and evaluate the initial efficacy and safety of Clomastine fumarate in the treatment of Williams syndrome.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the initial efficacy and safety of Clomastine fumarate in the treatment of Williams syndrome. The secondary objective is to study Clomastine fumarate in relation to mechanisms of action, safety, and/or pathological mechanisms. This study was an open-label study with a randomized, cross-over, placebo-controlled design. Each participant will be randomly assigned to two groups through baseline assessment (see study results), with Group A receiving the FDA-approved drug Clemastine at a weight-dependent dose (see dosing table below) for the first cycle and placebo for the second cycle. Group B will be treated with placebo for the first cycle and the FDA-approved drug Clemastine for the second cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Age 3-6 years old;
2. Positive fluorescence in situ hybridization (FISH) test confirmed Williams syndrome;
3. GTF2I gene mutation was detected by whole exon;
4. Heart safety variables are normal (e.g. normal ECG, blood pressure 120-129/80-84)

Exclusion Criteria:

1. WS patients with other gene mutations;
2. Used antihistamines, monoamine oxidase inhibitors, barbiturates and sedatives, as well as drugs affecting cognitive behavior, limb movement, white matter myelin, and MRI within 2 months before enrollment;
3. Patients with narrow-angle glaucoma, narrow peptic ulcer, pyloroduodenal obstruction, symptomatic prostatic hypertrophy and bladder neck obstruction; Accompanied by severe immunodeficiency disease;
4. Allergic to Clomastine fumarate or other arylalkylamine antihistamines or any receptor;
5. According to the recent interpretation of MRI and neuroradiology experts or WS, there are obvious brain lesions that are not related to WS disease;
6. Clinically significant metabolic, hematological, liver, immune, urinary, endocrine, neurological, pulmonary, psychiatric, skin, allergic, renal, or other major diseases that may affect the interpretation of study findings or patient safety in WS's judgment;

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-03-20 (Estimated); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anisotropy Score (FA) | baseline follow-up；second month；fourth month
  Measuring by Magnetic resonance diffusion tensor imaging (DTI)
Radial diffusion rate (RD) | baseline follow-up；second month；fourth month
  Measuring by Magnetic resonance diffusion tensor imaging (DTI)
Apparent dispersion coefficient（ADC） | baseline follow-up；second month；fourth month
  Measuring by Magnetic resonance diffusion tensor imaging (DTI)
Magnetization transfer ratio（MTR） | baseline follow-up；second month；fourth month
  Measuring by Magnetic resonance diffusion tensor imaging (DTI)
SRS Score 2(Social Response Scale2) score | baseline follow-up；second month；fourth month
  Assessing social skills
Peabody（Motion Estimation Timewarp）score | baseline follow-up；second month；fourth month
  Assessing motion skills
Gesell Development Scale | baseline follow-up；second month；fourth month
  Assessing neurodevelopment

SECONDARY OUTCOMES:
Differential pressure across valves | baseline follow-up；second month；fourth month
  Measuring by Cardiac color ultrasound
Thyroid hormone value | baseline follow-up；second month；fourth month
Conners Parent Symptoms Questionnaire Score | baseline follow-up；second month；fourth month
  Assessing adaptability
Vailand-3 scale | baseline follow-up；second month；fourth month
  Assessing neurodevelopment
CSHQ Children's Sleep Habits Questionnaire Score | baseline follow-up；second month；fourth month
  Assessing sleeping

CONTACTS AND LOCATIONS:
Overall Officials: cao aihua, post-doctoral, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Tainan, Shangdong, China

IPD SHARING:
Plan to Share IPD: No